CLINICAL TRIAL: NCT00203008
Title: A Survey to Assess the Incidence and Characteristics of Melanoma in Parkinson's Disease Patients
Brief Title: A Survey Study to See if Patients Diagnosed With Parkinson's Disease Have Higher Incidence of Melanoma
Status: Completed | Type: Observational
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: J. Michael Nicholas, PhD, Sr. Director, Teva Neuroscience
Other Study IDs: EP002
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2010-10-18 (Estimated); Status verified 2010-10

CONDITIONS: Parkinson's Disease; Malignant Melanoma
MeSH Terms: conditions — Parkinson Disease; Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Observational procedure: Patients will be examined and any suspicious skin abnormalities will be biopsied

SUMMARY:
Patients with Parkinson's disease will be seen by a dermatologist who will biopsy any suspicious skin lesions.

ELIGIBILITY:
Inclusion Criteria:

Confirmed diagnosis Parkinson's disease Patient able and willing to give informed consent Patient must not be taking any investigational drug at the time of enrollment

Exclusion Criteria:

unconfirmed, undocumented Parkinson's disease unable to give consent taking any investigational product

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients known to have Parkinson's Disease will be invited to join the study by their treating physicians as long as they are not taking investigational product.
Sampling Method: Non-Probability Sample
Enrollment: 2106 (Actual)
Dates: Start 2003-01; Study Completion 2003-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Schwartz, Ph.D., Study Director — Teva Neuroscience, Inc.